CLINICAL TRIAL: NCT01335100
Title: Does Botulinum Toxin Injections Improve Outdoor Activity in Children With Cerebral Palsy?- a Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Hilla Ben Pazi, MD, Shaare Zedek Medical Center
Other Study IDs: BTX-GPS
Record Dates: First submitted 2010-06-06; First posted 2011-04-14 (Estimated); Last update posted 2011-05-03 (Estimated); Status verified 2011-05

CONDITIONS: Cerebral Palsy
Keywords: Functional outcome; Quality of life; Global Positioning System (GPS); Advanced tracking technologies; Time-space activity.; walking speed; distances; number of walking events and destinations
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- ambulatory CP: ambulatory children with cerebral palsy undergoing Botulinum toxin injections to lower limbs
- controls: age and gender matched sibilings

SUMMARY:
Background:

Motor impairment limits social and recreational activities in children with cerebral palsy (CP), compromising participation and impacting on quality of life. Improvement of motor function by medical treatment may advance in participation of outdoor activities and expand social and recreational activities. While Botulinum toxin (BTX) injections are effective and safe treatment for spasticity in children with CP, there is insufficient evidence for improvement of motor function and enhanced participation in this population.

Objective:

To examine outdoor activity as a functional outcome following lower limb BTX in children with CP.

Methods:

In this pilot study the investigators will use Global Positioning Systems (GPS) to measure walking speed, distances, number of walking events and destinations in ambulatory children with CP following BTX injection to the lower limbs; age and gender matched sibling will be studied as a control group. Outdoor activity will be measured at 1, 3 and 6 months following BTX treatment will be compared to baseline and to those of siblings. Outdoor activity will be correlated with leisure activity preferences and quality of life questionnaires.

Significance: Improvement in outdoor activity following BTX injections in this pilot study will assist construction of a larger study evaluating participation and quality of life in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory children with CP following BTX injection to the lower limbs

Exclusion Criteria:

* significant psychomotor retardation, psychiatric symptoms or behavioral problem that may impact on outdoor activity prefernces

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: ambulatory children with CP following BTX injection to the lower limbs
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-03

PRIMARY OUTCOMES:
outdoor activity | 9 months

SECONDARY OUTCOMES:
leisure activity preferences and quality of life | 9 months for the pilot

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel